CLINICAL TRIAL: NCT00543335
Title: Phase I Trial of Sorafenib With Concurrent Thoracic Radiotherapy for Poor Prognosis Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Sorafenib and Thoracic Radiation for Patients With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0352; NCI-2010-00795 (Registry Identifier: NCI CTRP); NCT01636921 (obsolete NCT alias)
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; NSCLC; Radiation Therapy; Sorafenib; BAY 43-9006; Thoracic Radiation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib + Radiation Therapy (Experimental): Sorafenib starting dose 200 mg orally daily + 45 Gy total in 15 radiation treatments: 3 Gy per day, 5 days a week for 3 weeks
  Interventions: Drug: Sorafenib; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Sorafenib — Starting dose 200 mg PO (by mouth) Daily
  Other Names: BAY 43-9006
Procedure: Radiation Therapy — 45 Gy total in 15 radiation treatments: 3 Gy per day, 5 days a week for 3 weeks
  Other Names: RT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of sorafenib that can be given in combination with radiation therapy to people with lung cancer. The ability of both the study drug and radiation to control the disease will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Sorafenib is designed to block the function of important proteins in cancer cells. These proteins, when active, are in part responsible for the growth and behavior of cancer cells.

Study Drug Dose Escalation:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 4 groups of 3-6 participants will be enrolled in the Phase I portion of the study.

Enrolled in the Phase I portion, the dose of sorafenib you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of sorafenib. Each new group will receive a higher dose of sorafenib than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of sorafenib is found.

All participants will receive the same type and amount of radiation.

Study Drug Administration:

You will take sorafenib capsules 1-2 times every day beginning on Day 1 of radiation therapy. If you are in the first group on study, you will take the study drug 1 time. If you are in any other groups, you will take the study drug 2 times a day. You will take the study drug without food (1 hour before or 2 hours after eating).

Radiation Therapy:

Before receiving radiation therapy, you will have a "marking session". At this visit, you will have a computed tomography (CT) scan that will be used to help to plan out the radiation therapy. This will take about 45 minutes.

Before receiving radiation, you will also have a single photon computed tomography (SPECT) scan of your lungs.

You will be given 15 radiation treatments, once a day, 5 days a week, Monday-Friday. Each treatment will take about 30 minutes. You will sign a separate consent form for radiation therapy and the procedure will be described to you in more detail.

Clinical Visits:

You will have routine clinical visits every week while receiving radiation therapy. The information collected during these clinical visit will be used for the study. At these visits, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your blood pressure and weight.
* You will be asked about any side effects you may be experiencing and any new drugs you may be taking.
* You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation)
* Blood (about 3-4 teaspoons) will be drawn for routine tests.
* You will have any tests that doctor feels medically necessary

Urine will be collected every week while you are taking sorafenib and receiving radiation therapy for routine tests.

Length of Study:

You will remain on study for 6 weeks after you complete radiation therapy. You will be taken off the study early if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

You will have an end-of-study visit 4-6 weeks after you stop receiving radiation. At this visit, you will have a CT scan to check the status of the disease.

Follow-Up Visits:

Your first follow-up visit will be at 6 weeks (+/- 7 days) after radiation therapy and the second follow-up appointment will be at 10 weeks (+/- 7 days) after radiation therapy. You will then have follow up visits every 3 months. At these visits, you will go though the following:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your weight and blood pressure.
* You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation).
* You will be asked about any drugs you may be taking.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests.
* You will also have chest x-ray.
* You will have a computed tomography (CT) scan of your chest area.
* The location, type, and size of all measurable lesions will be recorded.
* If your doctor thinks it is necessary, you will have a positron emission tomography(PET)/CT scan.
* If your doctor thinks it is necessary, you will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart).
* You may have a lung perfusion scan to see if all regions of your lung are equally functional or not. This is called lung SPECT scan.
* You will have a lung functional test (PFT) if your doctor thinks it is necessary.

All these tests are routine examinations as you would have without participating in this study in order to know the status of the disease.

This is an investigational study. Sorafenib is FDA approved and commercially available for renal cell carcinoma. The radiation therapy schedule used for this study is standard treatment for lung cancer patients. The use of sorafenib with radiation therapy is investigational.

Up to 64 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven previously untreated or systemically treated poor prognosis NSCLC patients for whom palliative thoracic irradiation is the treatment of choice per standard of care.
2. Patients for whom palliative thoracic irradiation therapy to 45 Gy/15 FX is the recommended treatment by their treating radiation oncologist.
3. The primary tumor and/or regional lymphatic metastases must be evaluable radiographically.
4. Age >/= 18 years or older.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 or greater, weight loss </= 30% or less.
6. No prior radiation to the thorax.
7. Adequate bone marrow, liver and renal function as assessed by the following: * Hemoglobin >/= 9.0 g/dl * Absolute neutrophil count (ANC) >/=1,000/mm^3 *Platelet count >/ =100,000/mm^3 * Total bilirubin </= 1.5 times ULN or greater * ALT and AST </= 2.5 times the ULN (</= 5 * ULN for patients with liver involvement) * Creatinine </= 1.5 * ULN
8. Patients with distant metastasis are eligible.
9. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
10. Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
11. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
12. INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
13. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of M.D. Anderson Cancer Center. The only approved consent form is attached to this protocol.

Exclusion Criteria:

1. Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
2. Known hemorrhagic brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude hemorrhagic brain metastasis.
3. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
4. Uncontrolled hypertension defined as systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
5. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
6. Active clinically serious infection > CTCAE Grade 3.
7. Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
8. Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
9. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
10. Serious non-healing wound, ulcer, or bone fracture.
11. Evidence or history of bleeding diathesis or coagulopathy
12. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
13. Current use of St. John's Wort or rifampin (rifampicin).
14. Known or suspected allergy to sorafenib.
15. Any malabsorption problem.
16. Patients with squamous cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01-25 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) of sorafenib concurrent with thoracic radiation for poor prognosis NSCLC (phase I) | Continual reassessment of safety throughout study and determination of dose-limiting toxicities during and at end of 3 week cycles.

SECONDARY OUTCOMES:
Efficacy of combination assessed by tumor response and local progression failure (phase II) | 6 Months and 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD . Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org